CLINICAL TRIAL: NCT02360137
Title: Atherosclerotic Plaque Characteristics Associated With a Progression Rate of the Plaque and a Risk of Stroke in Patients With the carotId Bifurcation Plaque Study
Brief Title: Atherosclerotic Plaque Characteristics Associated With a Progression Rate of the Plaque in Carotids and a Risk of Stroke
Acronym: ANTIQUE
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital Ostrava (Other)
Collaborators: General Teaching Hospital, Prague (Other); Charles University, Czech Republic (Other); Palacky University (Other); Military University Hospital, Prague (Other); University of Ostrava (Other); Masaryk Hospital Usti nad Labem (Other); University Hospital Hradec Kralove (Other); Na Homolce Hospital (Other); University Hospital Olomouc (Other)
Responsible Party: Sponsor
Other Study IDs: 15-29410A
Record Dates: First submitted 2015-01-26; First posted 2015-02-10 (Estimated); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Carotid Artery Plaque
Keywords: carotids; plaque; characteristics; stroke
MeSH Terms: conditions — Carotid Stenosis; Plaque, Amyloid; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — atherosclerotic plaque
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with carotid plaque: Patients with carotid plaque treated using only drugs
- Patients with carotid stenosis: Patients with carotid stenosis indicated to carotid endarterectomy

SUMMARY:
Atherosclerosis is the most common cause of stroke. The aims of the project are to compare the visual and digital analysis of sonographic images of atherosclerotic plaque in carotids in vivo, in vitro and with a histological composition of the plaque obtained from patients indicated to carotid endarterectomy, to compare the characteristics of symptomatic and asymptomatic atherosclerotic plaques and, subsequently to verify a hypothesis that ultrasound can identify the sonographic plaque characteristics associated with an increased risk of plaque progression and of ischemic stroke (unstable plaque) in patients with carotid atherosclerosis. Identifying of the sonographic characteristics of unstable plaque will allow to improve indication criteria for carotid endarterectomy or stenting and also potential changing of a drug therapy in patients with unstable plaque in the future. Cost efficiency and availability of duplex ultrasound equipment may enable to improve diagnosis of unstable plaque using this new plaque characteristics evaluation in the majority of patients with carotid plaques.

DETAILED DESCRIPTION:
Objectives and aims The objective of the project is to identify measurable features of atherosclerotic plaque in carotids associated with plaque progression and increased stroke/TIA risk using duplex sonography and digital B-mode image analysis.

The project aims

1. to identify characteristics of carotic atherosclerotic plaque in ultrasound B-mode associated with a risk of progression or stroke/TIA onset - the "vulnerable" atherosclerotic plaque using

   1. visual assessment
   2. digital image analysis using a computer program
2. to determine the correlation of the ultrasound finding of carotic atherosclerotic plaque in a B-mode in vivo (before endarterectomy) and subsequently in vitro (after endarterectomy) in patients indicated to carotid endarterectomy using

   1. visual assessment
   2. digital image analysis using a computer program
3. to assess a correlation between histological evaluation of composition of atherosclerotic plaque obtained during carotid endarterectomy and ultrasound image of atherosclerotic plaque in a B-mode in vitro using

   1. visual assessment
   2. digital image analysis using a computer program
4. to compare histological and ultrasound findings in vitro and in vivo between asymptomatic and symptomatic atherosclerotic plaques in the carotid bifurcation using

   1. visual assessment
   2. digital image analysis using a computer program
5. to compare the features of asymptomatic and symptomatic atherosclerotic plaque in the carotid bifurcation using

   1. sonographic perfusion examination of plaque in vivo (after application of echocontrast agent)
   2. elastography

The grant project is in concordance with the scope, expected benefits, key objective of the Programme "Ensuring internationally comparable levels of healthcare research and use the results to improve the health of Czech population and to secure the current needs of the health sector in the Czech Republic" and the sub-objective 1.2.2. "The development of early diagnosis of cardiovascular and cerebrovascular disease and finding treatment modalities and procedures in the treatment of cardiovascular and cerebrovascular disease with greater therapeutic efficiency and greater parsimony for the patient."

Project design

1. Patients The project period will take 132 months. Total of 1863 patients with atherosclerotic plaques in the carotid bifurcation and internal carotid artery causing arterial stenosis ≥ 30% detected by duplex sonography will be included to the study. Patients indicated for carotid intervention according to the currently valid guidelines (American Heart Association/American Stroke Association [AHA], European Stroke Organisation [ESO]) will undergo carotid endarterectomy or carotid stenting. Patients will be screened and enrolled in sonographic laboratories of the Military University Hospital in Prague, Na Homolce Hospital Prague, University Hospital Ostrava, Olomouc and Hradec Kralove.

   Inclusion criteria: 1/ age 30 - 90 years, 2/ sufficient image quality of atherosclerotic plaque in the carotid bifurcation and ICA using ultrasound, 3/ independency of the patient (0 - 2 points in the modified Rankin scale), 4/ signed informed consent.

   Exclusion criteria: 1/ serious disease with a low probability of survival of at least 3 years, 2/ other objective obstacles preventing regular 6-month ultrasound scan.

   Clinical examination: Physical and neurological examinations and examinations of carotid arteries by duplex sonography will be performed in all patients at baseline and every 6 months for 3 years.
2. Sample size calculation The sample size for prospective follow-up of atherosclerotic plaques was based on an expected 5% difference in stroke risk between plaque characteristics. Pre-study calculations showed that a minimum of 1863 patients were needed to reach a significant difference with an alpha value of 0.05 (two-tailed) and a beta value of 0.8 assuming that 20 % of subjects will lost to follow-up.

   The sample size for patients undergoing carotid endarterectomy with subsequent in vitro sonographic and histological evaluation of atherosclerotic plaques was based on an expected Spearman's correlation coefficient ≥ 0.3 between histological and sonographic evaluation of atherosclerotic plaque (visual and digital image analysis). Pre-study calculations showed that a minimum of 152 patients were needed to reach a significant difference with an alpha value of 0.01 (after Bonferroni correction for 5 evaluated factors) and a beta value of 0.8 assuming that 20 % of plaques will not be suitable for evaluation.
3. Duplex sonographic examination of carotid arteries Standard duplex sonography of cervical vessels focusing on the carotid bifurcation and proximal part of the ICA with measurement of the maximum width of atherosclerotic plaque and transcranial duplex color-coded sonography will be performed in all all patients at baseline and thereafter in 6-month period for 3 years (totally 7 examinations). Examinations will be performed using high-end duplex ultrasound system ESAOTE MyLab Twice (ESAOTE, Genova, Italy) with linear probe LA435 (10 - 18 MHz), vascular preset, scanning depth 4.0 cm, 2 focuses in 2.0 and 3.0 cm; for transcranial duplex sonography, a phase array PA 240 (2 - 4 MHz) will be used. Free hand sonographic scanning will be performed in B-mode in longitudinal and transversal planes (continuous hand moving without changes of probe angle). Video sequences from both longitudinal and transversal scanning and images of cross-section of the plaque in subsequent distance of 0.5 mm will be saved and encoded. Visual characteristics of the plaque (echogenicity, homogeneity, surface, etc.) and digital image analysis using B-mode Assist System will be performed from each video sequence and each cross-section of the plaque. Sonographic examination of plaque perfusion in vivo after application of echocontrast agent (SonoVue, Bracco, Italy) and elastography will be performed in at least 25 patients.
4. Carotid endarterectomy Surgery will be undertaken according to standard protocols using general anesthesia in all patients at both centers (with > 400 carotid endarterectomies carried out during the last 5 years). All patients will be on uninterrupted long-term acetylsalicylic acid therapy (100 mg/day) or dual antiplatelat therapy during the perioperative period. A dose of 100 IU per 1 kg of body weight of unfractionated heparin (Heparin Léčiva, Zentiva, k.s., Prague, Czech Republic) will be administered routinely at least 3 - 5 min before flow arrest in carotid artery. The plaque in carotid bifurcation and proximal part of the ICA will be removed as a 1 block from the artery. Protamin (Protamin Meda-Ampullen, Legacy Pharmaceuticals Switzerland GmbH, Birsfelden, Switzerland) in a dose of 1 mL per 2,000 IU of unfractionated heparin will be administered 5 min after flow restoration in the ICA when needed. Clopidogrel (Trombex 75 mg, Zentiva, k.s., Prague, Czech Republic) will be administered 5 days after surgery (75 mg/day) when indicated.
5. Sonographic examination of atherosclerotic plaque in vitro All atherosclerotic plaques obtained during endarterectomy as a 1 block will be examined sonographically in vitro. Examination will be performed using the high-end duplex ultrasound system ESAOTE MyLab Twice (ESAOTE, Genova, Italy) with linear probe LA435 (10-18 MHz), vascular preset, scanning depth 2.0 cm, 2 focuses in 1.0 and 2.0 cm. Atherosclerotic plaques extracted from carotid arteries will be transported in a box with formaldehyde. Each plaque will be inserted to the open plastic box filled by HAES 130/04 Voluven solution (colloid plasma expander). Free hand sonographic scanning will be performed in B-mode in longitudinal and transversal planes (continuous hand moving without changes of probe angle). Video sequences from both longitudinal and transversal scanning and images of cross-section of the plaque in subsequent distance of 0.5 mm will be saved and encoded. Visual characteristics of the plaque (echogenicity, homogeneity, surface, etc.) and digital image analysis using B-mode Assist System will be performed from each video sequence and each cross-section of the plaque.
6. Histological processing and analysis of atherosclerotic plaque All atherosclerotic plaques obtained during endarterectomy as a 1 block will be processed and analysed histologically after sonographic examination. Visual characteristics of the plaque and digital image analysis using B-mode Assist System will be performed from each cross-section of the plaque.

ELIGIBILITY:
Inclusion Criteria:

* age 30 - 90 years
* sufficient image quality of atherosclerotic plaque in the carotid bifurcation and ICA using ultrasound
* independency of the patient (0 - 2 points in the modified Rankin scale)
* signed informed consent.

Exclusion Criteria:

* serious disease with a low probability of survival of at least 3 years
* other objective obstacles preventing regular 6-month ultrasound scan.

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The project period will take 54 months. Total of 413 patients with atherosclerotic plaques in the carotid bifurcation and internal carotid artery causing arterial stenosis ≥ 30% detected by duplex sonography will be included to the study - 152 patients indicated for carotid endarterectomy according to the currently valid guidelines (American Heart Association/American Stroke Association [AHA], European Stroke Organisation [ESO]) and 261 patients indicated for conservative treatment. Patients will be screened and enrolled in sonographic laboratories of the Military University Hospital in Prague and University Hospital Ostrava.
Sampling Method: Probability Sample
Enrollment: 1863 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Plaque progression | 10 years
  Sonographic and histological characteristics associated with plaque progression

SECONDARY OUTCOMES:
Stroke risk | 10 years
  Sonographic and histological characteristics associated with stroke or TIA risks, such as homogeneity, composition, echogenity index, plaque surface type
Mortality | 10 years
  Sonographic and histological characteristics associated with mortality, such as homogeneity, composition, echogenity index, plaque surface type
Sonographic plaque characteristics correlation | 1 year
  Sonographic plaque characteristics correlation, using Spearman correlation coefficient to verify the existence of correlations between carotid atherosclerotic plaque in a B-mode in vivo (before endarterectomy) and subsequently in a B-mode in vitro (after endarterectomy) in homogeneity, composition, echogenity index, plaque surface type
Histological and sonographic plaque characteristics correlation | 1 year
  Histological and sonographic plaque characteristics correlation, using Spearman correlation coefficient to verify the existence of correlations between variables - homogeneity, composition, echogenity index, plaque surface type

CONTACTS AND LOCATIONS:
Overall Officials: David Skoloudík, MD, Prof, Study Chair — University Hospital Ostrava
Locations (1):
- University Hospital Ostrava, Ostrava, Czech Republic, Czechia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Pakizer D, Salounova D, Skoloudik D. Extracranial carotid plaque calcification and its association with risk factors for cerebrovascular events: insights from the ANTIQUE study. Front Neurol. 2025 Jan 29;16:1532883. doi: 10.3389/fneur.2025.1532883. eCollection 2025. PMID 39944551
- [Derived] Skoloudik D, Kesnerova P, Hrbac T, Netuka D, Vomacka J, Langova K, Herzig R, Belsan T. Risk factors for carotid plaque progression after optimising the risk factor treatment: substudy results of the Atherosclerotic Plaque Characteristics Associated with a Progression Rate of the Plaque and a Risk of Stroke in Patients with the carotid Bifurcation Plaque Study (ANTIQUE). Stroke Vasc Neurol. 2022 Apr;7(2):132-139. doi: 10.1136/svn-2021-001068. Epub 2021 Dec 1. PMID 34853082
- [Derived] Fadrna T, Miksova Z, Herzig R, Langova K, Licman L, Skoloudik D. Factors influencing quality of life in patients followed in the neurosonology laboratory for carotid stenosis. Health Qual Life Outcomes. 2018 Apr 27;16(1):79. doi: 10.1186/s12955-018-0902-2. PMID 29703211